CLINICAL TRIAL: NCT06603454
Title: Preoperative Chest CT-imaging in Surgical Aortic Valve Replacement with or Without CABG: a Randomized Controlled Trial
Brief Title: Preoperative Chest CT-imaging in Surgical Aortic Valve Replacement with or Without CABG
Acronym: GUIDE-SAVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Romy Hegeman (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor-Investigator, Romy Hegeman, Research Coordinator, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL77700.100.21
Record Dates: First submitted 2024-07-27; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative CT (Active Comparator): Contrast-enhanced computed tomography of the aorta including the femoral arteries.
  Interventions: Radiation: Preoperative CT
- No preoperative CT (No Intervention)

INTERVENTIONS:
Radiation: Preoperative CT — Preoperative contrast enhanced CT
  Arms: Preoperative CT

SUMMARY:
Rationale When determining the strategy for aortic valve replacement, echocardiography is still considered the golden standard (1). While pre-procedural MSCT is standard of care in TAVR patients, this is not yet part of routine clinical practice in SAVR patients. The researchers hypothesise that when atherosclerosis of the ascending aorta is identified preoperatively on contrast-enhanced multi-slice computed tomography (MSCT), the subclinical perioperative stroke rate (as detected on diffusion-weighted magnetic resonance imaging (DW-MRI)) can be reduced by modification of the operative strategy if necessary.

DETAILED DESCRIPTION:
When determining the strategy for aortic valve replacement, echocardiography is still considered the golden standard (1). While pre-procedural MSCT is standard of care in TAVR patients, this is not yet part of routine clinical practice in SAVR patients. The investigators hypothesise that when atherosclerosis of the ascending aorta is identified preoperatively on contrast-enhanced multi-slice computed tomography (MSCT), the subclinical perioperative stroke rate (as detected on diffusion-weighted magnetic resonance imaging (DW-MRI)) can be reduced by modification of the operative strategy if necessary.

The primary objective is to assess whether the use of pre-operative MSCT will reduce subclinical stroke rates (i.e., ischemic brain lesions) as identified with the use of DW-MRI after SAVR with or without concomitant CABG surgery.

The secondary objective is to assess whether the use of pre-operative MSCT will improve neurological assessment score, reduce clinical stroke, mortality, change in intervention strategy (pre- or intra-operatively), cannulation strategy and clamping strategy as well as reduce procedural times and improve quality of life (with the application of EQ-5D and KCCQ questionnaires).

This is a prospective, multicenter, parallel, open-label randomized controlled trial (RCT) with a 1:1 randomization including patients aged 18 years and older accepted for SAVR with or without concomitant CABG by the Heart Team at the St. Antonius Hospital Nieuwegein. All patients enrolled in the study will be randomized to additional pre-operative MSCT or no additional pre-operative MSCT. Postoperatively, a DW-MRI will be made in all patients. The trial will end after 30-day follow-up of all enrolled patients.

The main primary endpoint is the incidence of subclinical stroke rate (i.e., presence of new ischemic brain lesions) as identified with the use of DW-MRI made within one week postoperatively or before discharge. Secondary endpoints include the National Institutes of Health Stroke Scale (NIHSS) score within one week postoperatively (targeted at day two postoperatively), clinical ischemic stroke (conform VARC-3),transient ischemic attack diagnosed by a neurologist within one week postoperatively, defined by transient focal neurological signs or symptoms lasting < 24 h presumed to be due to focal brain, spinal cord or retinal ischemia, but without evidence of acute infarction by neuroimaging or pathology, or with no imaging performed (conform VARC-3), mortality at discharge (normally at three to five days postoperatively) or within one week postoperatively (if discharge is > 1 week postoperatively) and at three months postoperatively, the change in intervention strategy, the change in cannulation strategy, the change in clamping strategy, procedural times and the quality of life at three months postoperatively (assessed by EQ-5D and KCCQ)

When severe calcification of the ascending aorta is identified preoperatively on multi-slice computed tomography (MSCT), the operative strategy can be modified if necessary. This could possibly prevent stroke or even mortality in the study patients randomized to additional pre-operative MSCT. The MSCT will take 5-10 minutes. Only low-dose contrast-enhanced CT will be used, which results in a very low radiation risk. With application of too high dosages of contrast, there is a slight chance of kidney insufficiency. Furthermore, an allergic reaction to contrast could occur. However, patients with known allergies to contrast and patients with low renal function will be excluded from participation in this trial.

The patients receiving a preoperative CT-scan will have to be informed about all incidental findings found on the CT-scan. A possible disadvantage is found in the additional costs of a CT-scan, but the costs associated with stroke would outweigh the costs of a preoperative CT-scan. All patients will receive a DW-MRI before discharge. Contra-indications for MRI include pacemaker wires or implantable cardioverter defibrillators (ICDs), metallic implants, cochlear/ear implants, Swan-Ganz catheter, claustrophobia and contrast allergy. The presence of an aortic valve prosthesis is not a contra-indication for DW-MRI scanning.

All patients will be asked to fill out a questionnaire at baseline and within 90 days postoperatively. Since this will soon be implemented as part of standard care, the latter is not seen as extra burden for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary symptomatic severe aortic valve stenosis (defined as an aortic valve area of <1.0cm2 and either a mean valve gradient of at least 40mmHg or a peak velocity of at least 4.0 m/s)
* Accepted for SAVR (either planned to be done by a limited access approach (partial J-shaped sternotomy or right anterior thoracotomy or conventional median sternotomy approach at the preference of the patient and/or the discretion of the surgeon) with or without concomitant CABG by the Heart Team
* Informed consent

Exclusion Criteria:

* Previous aortic valve replacement
* Emergency procedure
* Pregnant women
* Renal failure (eGFR <30 ml/min.)
* Known contrast allergy
* Patient unwilling to be informed about unrequested findings on the CT scan or DW-MRI scan
* Contra-indication for MRI (e.g. permanent pacemaker or ICD that can not be inactivated per order of the pacemaker or ICD technician, morphine or insulin pump, neurostimulator). All patients will fill out a MRI checklist to additionally check for (new) safety contra-indications for MRI.
* Patient who did not agree to the informed consent and/or refused to participate
* Patient unable to understand the informed consent/study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Subclinical stroke rate | Within 90 days post procedure
  Subclinical stroke rate (i.e., presence of new ischemic brain lesions) as identified with the use of DW-MRI made within one week postoperatively or before discharge (in case of prolonged ICU stay).

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale | within one week postoperatively (targeted at day two postoperatively)
  National Institutes of Health Stroke Scale, ranging 0 - 42. Higher scores refer to a more severe stroke.
Clinical ischemic stroke (conform VARC-3) | Within one week postoperatively
  The incidence of clinical ischemic stroke (conform VARC-3) diagnosed by a neurologist within one week postoperatively, defined by the acute onset of focal neurological signs or symptoms conforming to a focal or multifocal vascular territory within the brain, spinal cord or retina and fulfilling one of the following criteria:
  * Signs or symptoms lasting ≥24 h or until death, with pathology or neuroimaging evidence of CNS infarction, or absence of other apparent causes
  * Symptoms lasting < 24 h, with pathology or neuroimaging evidence of CNS infarction in the corresponding vascular territory
TIA diagnosed by a neurologist | One week postoperatively
  The incidence of TIA diagnosed by a neurologist within one week postoperatively, defined by transient focal neurological signs or symptoms lasting < 24 h presumed to be due to focal brain, spinal cord or retinal ischemia, but without evidence of acute infarction by neuroimaging or pathology, or with no imaging performed (conform VARC-3).
Change in intervention strategy | After hospital admission but before the end of surgery
  Change in intervention strategy (no unfavourable change, cancellation of surgery, switch to TAVR preprocedural, conversion from limited access to conventional full median sternotomy, conversion to TAVR)
Change in cannulation strategy | During procedure
  Change in cannulation strategy (no change, use of different cannula, avoiding cannulation of the ascending aorta/arch (thus femoral or subclavian cannulation), higher cannulation (arch), lower cannulation, echo-guided cannulation)
Change in clamping strategy | During procedure
  Change in clamping strategy (no change, change of clamping site, no clamping)
Procedural times | During procedure
  Implantation time (defined period from start of the first suture until the completion of the prosthesis implantation = fixation of last suture), surgical time, aortic cross-clamp (ACC) time, cardio-pulmonary bypass (CPB) time. All times in minutes.
Quality of life at three months postoperatively (assessed by EQ-5D and KCCQ) | At baseline (prior to procedure) and 90 days post procedure
  All scores are represented on a 0-to-100-point scale. Higher score refers to preferabel outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Klein, MD, PhD, Principal Investigator — St. Antonius Hospital; Prof. Jurriën C ten Berg, MD, PhD, Principal Investigator — St. Antonius Hospital; Martin C Swaans, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Hospital, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
IPD data can be shared upon reasonable request to the corresponding author.